CLINICAL TRIAL: NCT06824363
Title: Proof of Principle Study Evaluating Single Dose Dual Immune Checkpoint Inhibitors to Increase Intra-tumoral T Cells in Esophageal, Gastroesophageal Junction, and Gastric Adenocarcinomas With ARID1A Mutations: ESR-22-22082
Brief Title: ProofPrincip IntraTu TCells SinglDoseImmunCheckpoinInhib Gastro-Esophage Adenocarcinoma w/ARID1a Mu
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Farshid Dayyani, HS Associate Clinical Professor, Department of Medicine, Division of Hematology, Oncology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6069; UCI 23-173 (Other: UCI CFCCC)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult; Malignant Solid Tumor; Stomach Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tremelimumab and Durvalumab (Experimental): Tremelimumab 300 mg IV, single-dose, day 1 Durvalumab 1500mg IV, single-dose, day 1
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tremelimumab — single dose, 300mg IV, day 1
Drug: Durvalumab — single dose, 1500 mg IV, day 1

SUMMARY:
This is a proof of principle clinical trial determining efficacy of single dose dualimmune checkpoint inhibitors to increase intra-tumoral T cells in esophageal, gastroesophageal junction, and gastric adenocarcinomas. These are subjects who have not previously been treated for their disease, who are willing to undergo biopsy procedures, who's disease has not spread to other parts of the body, who's tumors have ARID1A mutations.

ELIGIBILITY:
Inclusion Criteria:

* Non metastatic GEC including locally advanced unresectable
* Treatment naïve
* Histologically proven adenocarcinoma of the esophagus or the stomach with ARID1a mutation either by liquid biopsy (ctDNA) or tissue NGS/WES
* MSI-Stable or pMMR
* Age ≥ 18 years
* Body weight > 66 pounds
* ECOG ≤ 2
* Repeat biopsy feasible
* No clinically significant autoimmune disease

Exclusion Criteria:

* Patients with known metastatic disease
* Prior systemic treatment for esophagus, GEJ, or the stomach adenocarcinoma
* Patients with uncontrolled autoimmune disease per investigator discretion
* Inability or refusal to undergo biopsy procedures to obtain tissue samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects Completing Study Treatment | 2 Years
  Percentage of Subjects Completing the Study Treatment
Percentage of Subjects Completing Post-Treatment Biopsy | 2 Years
  Percentage of Subjects Completing the Post-Treatment Biopsy

SECONDARY OUTCOMES:
Percent Change in the Proportion of Intra Tumoral Effector T-cells | 2 years
  Assessment of Effects on Tumor Microenvironment Composition based on the percent change in the proportion of intra tumoral effector T-cells (CD3/CD8) at 2-6 weeks post single dose of STRIDE regiment compared to that at baseline
Assessment of effects on circulating cytokines in a 96-cytokine-discovery assay. | 2 years
  Assessment of effects on circulating cytokine from whole blood collection at baseline and after receiving Tremelimumab and Durvalumab. Blood samples will be used to perform a 96-cytokine-discovery assay.
  https://www.evetechnologies.com/product/new-human-cytokine-chemokine-96-plex-discovery-assay-array-hd96/
Number of Patients who received one dose of Tremelimumab and Durvalumab with reported Adverse Events | 2 years
  Evaluation of safety and adverse events of patients who received one dose of Tremelimumab and Durvalumab using the CTCAE version 5.0
Comparison of T-Cell Infiltration in Various Tumor Mutations | 2 years
  Comparison of T-Cell Infiltration in ARID1A mutated tomors to ARID1A wile-type tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States